CLINICAL TRIAL: NCT03399487
Title: An Open-label, Multicenter, Phase II Study of LDK378 in Patients With Non-small Cell Lung Cancer Harboring ROS1 Rearrangement
Brief Title: A Study of LDK378 in Patients With Non-small Cell Lung Cancer Harboring ROS1 Rearrangement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0240
Record Dates: First submitted 2017-09-21; First posted 2018-01-16 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Non-small Cell Lung Cancer Harboring ROS1 Rearrangement
Keywords: NSCLC; ROS1 rearrangement; Ceritinib; LDK378
MeSH Terms: interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): This study is a phase II, single-arm, open label study. All participating patients must sign on the written informed consent form, and a separate form of consent will be used for the use of tissue for the biomarker research.
  This clinical study is targeted for the patients who harbor ROS1 rearrangement and all patients will be treated with LDK378 750mg daily. The treatment period begins on Day 1 of Cycle 1 and 1 cycle consists of 28 days.
  Patients will be continued to receive study drug until the end of study unless the patients in disease progression, unacceptable toxicity, withdrawn consent, or by the investigator's judgment.
  Interventions: Drug: LDK378(Ceritinib)

INTERVENTIONS:
Drug: LDK378(Ceritinib) — This study is a phase II, single-arm, open label study. All participating patients must sign on the written informed consent form, and a separate form of consent will be used for the use of tissue for the biomarker research.
  This clinical study is targeted for the patients who harbor ROS1 rearrangement and all patients will be treated with LDK378 750mg daily. The treatment period begins on Day 1 of Cycle 1 and 1 cycle consists of 28 days.

SUMMARY:
Lung cancer is the most leading cause of cancer-related mortality worldwide. Most of the patients with lung cancer are advanced stage at the time of diagnosis.

The two oncogenes that are important in lung cancer are epidermal growth factor receptor (EGFR) and K-ras, mutated in 10% and 15% of non-small cell lung cancer (NSCLC) patients. Large-scale DNA sequencing efforts have identified mutations in BRAF, PI3KCA and ERBB2 that together represent another 5% of NSCLC patients. The success of EGFR tyrosine kinase inhibitors (TKIs), such as gefitinib or erlotinib, and more recently ALK/MET TKI, crizotinib, highlights the need to develop more genetically matched therapies. Therefore, genetic classification of lung cancer has become increasingly important along with the advances with targeted therapies.

ROS1 is a receptor tyrosine kinase with constitutive kinase activity. ROS1 was previously discovered in cell lines where ROS1 fused with other proteins to act as a driver oncogene. In 2007, Rikova et al reported ROS1 fusion as driver mutations in NSCLC cell line (HCC78; SLC34A2-ROS1) and NSCLC patient (CD74-ROS1). Li et al also found about 1% of samples harboring CD74-ROS1 fusion in 202 resected lung adenocarcinomas from never smokers. The incidence was as high as 10% in East Asian population. Currently there are now at least 13 ROS1 fusion variants involving 8 fusion partners (CD74-, SLC34A2-, FIG-, TPM3-, SDC4-, LRIG3-, ERZ-, KDERL2-) identified in ROS1 positive NSCLC.

Interestingly, preclinical and clinical data have shown ROS1-positive tumors are sensitive to crizotinib, because of potentially high common amino acid residues in the kinase domain between ALK and ROS1, which explain why crizotinib can inhibit both ROS1 and ALK to similar extent. Preliminary report from a phase I clinical trial of crizotinib in the ROS1-positive NSCLC expansion cohort showed an overall response rate (ORR) of 57%. Given that crizotinib has made remarkable clinical outcomes in phase I trial of ALK-positive NSCLC patients, clinical development of ROS1 inhibitors, including crizotinib, should be accelerated to provide targeted therapies to ROS1-positive NSCLC patients.

DETAILED DESCRIPTION:
Recently, our group found the prevalence of ROS1 rearrangement reached up to 3.2% in clinically selected population (never smokers) and 5% in genetically selected population (EGFR-/ALK-wild-type). These data strongly suggests that ROS1 rearrangement is a potential therapeutic target with relatively high incidence. In this study, investigator confirmed the presence of ROS1 fusion by RT-PCR and correlation between FISH and IHC (Cell Signaling Technology®).

LDK378 is an orally highly selective and potent ALK kinase inhibitor. In preclinical studies, LDK378 has much lower IC50 values than crizotinib in cell lines engineered to express ROS1 rearrangement (0.15 nM versus 3 nM) and is approximately 20-fold more potent. LDK378 is a potent inhibitor of tumor growth in rodent models of both ALCL and NSCLC.

Investigators suggest a phase II trial of LDK378 in advanced non-small cell lung cancer patients with ROS1 rearrangement. The aim of current trial is to evaluate the antitumor efficacy and safety profile of LDK378.

ELIGIBILITY:
Inclusion criteria

* histologically or cytologically confirmed, stage IV or recurrent NSCLC that carries a ROS1 rearrangement, as per anchored multiplex PCR
* ECOG performance status of 0 to 2
* Male or female≥ 20 years of age
* treatment naive or may be allowed up to 2 prior systemic anti-cancer therapy for their stage IV or recurrent NSCLC, which includes cytotoxic chemotherapy and I-O, but excludes crizotinib.
* measurable lesion (using RECIST 1.1 criteria)
* measurable lesion (using RECIST 1.1 criteria)
* archival tissue sample available, collected either at the time of diagnosis of NSCLC or any time since
* Subjects who meet the following criteria:

  * ANC 1.5 x 109/L -Platelet 100 x 109/L
  * creatinine 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) 3 x ULN (If there is Liver Metastasis 5 x ULN
  * Total bilirubin 1.5 x ULN
* written informed consent prior to any study specific procedures
* Leptomeningeal carcinomatosis may be included

Exclusion criteria

* More than two actionable mutations
* Patients who received prior crizotinib therapy
* Any major operation or irradiation within 4 weeks of baseline disease assessment
* Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
* Subjects with symptomatic central nervous system (CNS) metastases who are neurologically unstable or who have CNS complications that require urgent neurosurgical intervention(e.g. resection or shunt placement)
* Other co-existing malignancies or malignancies diagnosed within the last 3 years with the exception of basal cell carcinoma or cervical cancer in situ or treated thyroid cancer.
* Subjects with an uncontrolled major cardiovascular disease (including AMI within 12 months, unstable angina within 6 months, over NYHA class III congestive heart failure, congenital long QT syndrome, 2° or more AV Block and uncontrolled hypertension)
* Pregnant or lactating female
* Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention).
* Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with LDK378 and for the duration of participation (see Appendix 1 Tables):
* Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
* Strong inhibitors or strong inducers of CYP3A4/5 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
* Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, CYP2C8 and/or CYP2C9 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
* Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (eg, dabigatran, rivaroxaban, apixaban).
* Unstable or increasing doses of corticosteroids
* enzyme-inducing anticonvulsive agents
* herbal supplements
* Patients who have received thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs), radiotherapy ≤ 2 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study treatment is allowed.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
(ORR) overall response rate | 2 years
  The primary purpose is to investigate the overall response rate (ORR) of LDK378 by independent review committee (IRC) (Tumor assessment will measure the change of tumor size).

SECONDARY OUTCOMES:
PFS (progression-free survival ) in months | up to 2 years
  Progression-free survival in months
OS (overall survival) in months | up to 5 years
  Overall survival in months
DCR (disease control rate) in percentage | After study completion (an average of 2 year)
  Disease control rate in percentage
Incidence of Treatment-related adverse events in AE event name and grade | After study completion (an average of 2 year)
  Incidence of treatment-related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No